CLINICAL TRIAL: NCT04374942
Title: Protecting Frontline Health Care Workers From COVID-19 With Hydroxychloroquine Pre-exposure Prophylaxis: A Randomized, Placebo-controlled Multi-Site Trial in Toronto, Canada
Brief Title: Does Hydroxychloroquine Before & During Patient Exposure Protect Healthcare Workers From Coronavirus?
Acronym: HEROs
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to unproven issues associated with hydroxychloroquine use and safety, further complicated by media and political misinformation which in effect rendered all global studies on HCQ to stop enrolling participants.
Sponsor: Megan Landes (Other)
Responsible Party: Sponsor-Investigator, Megan Landes, Attending Physician, Emergency Department, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HEROs Protocol 1.5; ISRCTN14326006 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Pre-Exposure Prophylaxis; Coronavirus; SARS-CoV 2
Keywords: Hydroxychloroquine; PrEP; Pre-exposure Prophylaxis; COVID-19; Coronavirus; SARS-CoV 2
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: The HEROS study is a double-blind, randomized placebo controlled trial of oral HCQ 400 mg taken once daily for three months as PrEP to prevent COVID-19 in health care workers in the emergency department.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial is fully-blinded, at the level of the participant, study coordinator, and investigator. Study drug and placebo will be identical in appearance and will be provided by the manufacturer. They will be packaged in identical bottles and dispensed by the Research Clinical Trials Pharmacy at UHN.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study drug arm (Experimental): 50% of participants will be randomized to the study drug arm, and will take 400mg hydroxychloroquine orally once a day for three months (Day 1-90).
  Interventions: Drug: Hydroxychloroquine
- Placebo arm (Placebo Comparator): 50% of participants will be randomized to the placebo arm, and will take placebo orally once a day for three months (Day 1-90).
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydroxychloroquine — Oral Hydroxychloroquine, 400 mg taken once daily, for three months as pre-exposure prophylaxis to prevent COVID-19 in health care workers in the emergency department.
  Arms: Study drug arm
Drug: Placebo oral tablet — Placebo pill (same formula as Hydroxychloroquine without active ingredient) taken once daily, for three months.
  Arms: Placebo arm

SUMMARY:
On 11 March 2020, the World Health Organization declared SARS-CoV-2 (commonly called COVID-19) a global pandemic. As in any pandemic, maintaining the health and safety of the healthcare workforce is of great importance as health care workers (HCW) remain a critical line of defence against the spread of COVID-19 and play a vital role in the recovery of those already infected. Frontline HCW, such as those in the emergency department (ED), are at high risk of contracting COVID-19 due to their close proximity to patients who may have the virus. The impact of frontline HCW becoming ill and thus unable to go to work is equally high, and of grave risk to the function of the healthcare system and the ability to minimize the impact of the current pandemic. This study aims to evaluate whether hydroxychloroquine (HCQ), a well-tolerated drug typically used in the prevention of malaria transmission and rheumatic disease, taken before and during exposure to patients with COVID-19, is effective at reducing COVID-19 infections among ED health care workers.

DETAILED DESCRIPTION:
On March 11th, 2020, the World Health Organization (WHO) declared coronavirus disease (COVID-19) caused by severe acute respiratory virus coronavirus 2 (SARS-CoV-2) a pandemic. As of March 22, 2020 there have been over 267,013 confirmed cases and 11,201 deaths in 185 different countries or regions; it is quickly overwhelming health care systems worldwide to detrimental effect. Even with current moderate interventions imposed, estimates predict that 10-18% of the Canadian population will be infected with the virus by its peak in July. Health care workers (HCWs) remain a critical line of defence in the fight against this pandemic and maintaining their health is not only an important social responsibility of the government, but it is also of vital national interest to treat and control others infected with this virus or sick with other disease.

Estimates from China indicate that HCWs make up 3.8% of cases, while in Italy it is reported to be much higher - 8.3%. Early numbers from front-line workers in Italy suggested up to 20% of HCWs become infected with COVID-19, and these rates are approximately 3 times higher than the general population. When HCWs become sick, not only do they risk dying, but they also must take weeks away from work limiting the ability of the health care system to function. The fear associated with becoming ill also causes higher rates of missed work and higher rates of burnout, as seen with previous outbreaks. It is also now clear that asymptomatic transmission of COVID-19 not only occurs, but may even be the most important factor in spread of the virus. HCWs may therefore become vectors of viral spread to those who are the most vulnerable in other areas of the hospital. Preventing HCWs from acquiring SARS-CoV-2 should therefore be of the utmost importance to national interests.

Repurposing drugs already known to be safe and tolerable in humans provides a major advantage in a pandemic where time is critical. Of candidate drugs, chloroquine (CQ) and its derivative hydroxychloroquine (HCQ), have shown some promise. Originally an anti-malarial medication, CQ exerts direct antiviral effects by inhibiting pH-dependent steps of the replication of several viruses, including coronaviruses. It also has immunomodulatory effects, suppressing the release of TNFα and IL-6, which are involved in the inflammatory complications of several viral diseases. In vitro data has shown that CQ potently blocks virus infection at low micromolar concentrations with a high selectivity index. CQ is also widely distributed throughout the body, including the lungs, after oral administration. An early clinical trial of more than 100 COVID-19 patients in China reported that CQ was superior to placebo in inhibiting pneumonia, improving lung imaging, promoting viral seroconversion, and shortening the disease course, although data was not released. Based on those results experts in China recommended CQ 500mg twice daily for ten days in all patients with COVID-19. HCQ has also been shown to also have anti-SARS-CoV-2 activity in vitro and may actually be more potent. It has a better safety profile than CQ (during long term use), and allows a higher daily dose, with fewer concerns of drug-drug interactions. Preliminary clinical data also suggests that HCQ may lead to significantly faster viral clearance in COVID-19 patients as assessed by nasopharyngeal swab (70% vs. 12.5%, p=0.001).

Pre-exposure prophylaxis (PrEP) offers the ability to protect front-line HCWs from illness, decrease nosocomial spread of SARS-CoV-2, and prevent loss of work force due to illness. Rigorous testing of HCQ for this purpose is critical at this time. The investigators therefore aim to conduct the first randomized placebo-controlled trial of HCQ to prevent COVID-19 infections in emergency departments (ED) as they prepare for escalating rates of COVID-19 in Toronto, Canada.

ELIGIBILITY:
Inclusion Criteria:

* Health care worker (HCW) in the emergency department who is anticipated to work at least 10 shifts over the duration of the study period (minimum 6 hours per shift) and anticipated to remain in the emergency department for the duration of the study (i.e., not transferring to another unit). For the purposes of the study, "health care workers" are physicians (including residents), nurses, nurse practitioners, physician assistants, respiratory therapists, X-ray technicians, social workers and support staff (including but not limited to house-keeping, and porters).
* Age ≥18 years.
* Ability to communicate with study staff in English

Exclusion Criteria:

* Currently pregnant, planning to become pregnant during the study period, and/or breast feeding
* Known hypersensitivity/allergy to hydroxychloroquine or to 4-aminoquinoline compounds.
* Current use of hydroxychloroquine for the treatment of a medical condition.
* Known prolonged QT syndrome, or concomitant medications which simultaneously may prolong the QTC that cannot be temporarily suspended/replaced. These are including but not limited to Class IA, IC and III antiarrhythmics; certain antidepressants, antipsychotics, and anti-infectives; domperidone; 5-hydroxytryptamine (5-HT)3 receptor antagonists; kinase inhibitors; histone deacetylase inhibitors beta-2 adrenoceptor agonists.
* Known pre-existing retinopathy.
* Disclosure of self-administered use of hydroxychloroquine or chloroquine within 12 weeks prior to study. This window allows five half-lives of HCQ (i.e. 21 days) to pass before being reintroduced to the drug.
* Confirmed symptomatic COVID-19 at time of enrollment, i.e. symptom of COVID-19 at enrollment with confirmation of SARS-CoV-2 infection by viral detection as performed according to local guidelines for symptomatic HCWs. All participants with COVID-19 symptoms at enrollment will be directed to have confirmatory testing (within the department or occupational health as per the site guidelines). Participants who are negative for SARS-CoV-2 will be redirected to enrollment procedures; those testing positive will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Microbiologically confirmed COVID-19 (SARS-CoV-2 infection) | Samples collected at day 0, 30, 60, 90 and 120
  This is a composite endpoint which includes any positive result from a validated SARS-CoV-2 diagnostic assay including detection of viral RNA, or seroconversion by day 104 (14 days after end of the randomization period).

SECONDARY OUTCOMES:
Adverse events | Assessed at day 30, 60, 90, and day 120
  Assessed using the DAIDS Table for Grading the Severity of Adverse Events
Symptom duration of COVID-19 | Collected every 7 days from day 7 to day 120
  Collected weekly from participants via self-report, sent by email
Days of hospitalization attributable to COVID-19 | Collected every 7 days from day 7 to day 120
  The number of days (or partial days) spent admitted to an acute care hospital during the study period
Respiratory failure requiring ventilatory support attributable to COVID-19 | Collected every 7 days from day 7 to day 120
  the number of days (or partial days) requiring i) non-invasive and ii) endotracheal intubation with ventilation during the study period
Mortality | Collected every 7 days from day 7 to day 120
  Mortality attributable to COVID-19 and all-cause mortality during the study period
Impact on work eligibility | Collected every 7 days from day 7 to day 120
  Number of days ineligible/unable to work due to COVID-19
Seropositivity | Blood collected at day 0, 30, 60, 90, 120
  COVID-19 reactive serology
Short-term psychological impact | Measured at day 1, 60, 120
  Short-term psychological impact of exposure to COVID-19 measured using the K10, a validated measure of non-specific psychological distress, with a standard cutoff score of ≥16

CONTACTS AND LOCATIONS:
Overall Officials: Megan Landes, MD, Principal Investigator — University Health Network, Toronto; Kevin Kain, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
At the time of completion of the analysis of primary and secondary outcomes, the HEROS Steering Committee will review all applications for use of participant level data and make recommendations.